CLINICAL TRIAL: NCT04334785
Title: Evaluation for the Effectiveness and Safety of Cryo-ablation in the Treatment of Early Invasive Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N024
Record Dates: First submitted 2020-03-31; First posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- cryo-ablation group (Experimental): In the first stage, for patients who meet the criteria, cryo-ablation will be conducted for the lump of invasive breast cancer, and traditional surgery will be conducted within 32days after cryo-surgery. In the second stage, for patients who meet the criteria, cryo-ablation will be conducted, and 5-year effectiveness and safety will be evaluated subsequently.
  Interventions: Device: cryo-ablation

INTERVENTIONS:
Device: cryo-ablation — Under the guide of ultrasound, cryo-ablation for the lump of early invasive breast cancer will be conducted.

SUMMARY:
Recently, researchers in America reported a clinical research (Alliance Z1072) which proved that cryo-ablation could be considered as a non-surgical treatment of early-stage breast cancer. The long term effectiveness and safety of cryo-ablation in early invasive breast cancer is still unknown. Therefore, this prospective study are designed to evaluate the effectiveness and safety of cryo-ablation in early invasive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

stage 1:

1. female
2. ≥18 years old
3. invasive ductal carcinoma proved by core needle biopsy. Other type of breast cancer should be well considered and decided by investigators. Pathological report should be complete (with the result of ER, PR , HER2, KI67 etc., and FISH report of ERBB2 gene if necessary).
4. lump can be detected by ultrasound.
5. image results (including ultrasound, mammography and MR image) prove the lump is single-center, the maximum diameter of the lump <2cm.
6. with enough breast tissue, and enough space from lump to skin.
7. patients is not pregnant and has no plan for pregnancy in 2 years.
8. ECOG level: 0-2
9. serum creatinine≤1.1 mg/dl
10. for patients with double side (left and right side) breast cancer, both side of the tumor should meet the inclusion criteria.
11. patients are accessible for the follow up and mentally healthy.

stage 2:

1. female
2. ≥18 years old
3. invasive ductal carcinoma proved by core needle biopsy. Other type of breast cancer should be well considered and decided by investigators. Pathological report should be complete (with the result of ER, PR , HER2, KI67 etc., and FISH report of ERBB2 gene if necessary).
4. lump can be detected by ultrasound.
5. image results (including ultrasound, mammography and MR image) prove the lump is single-center, the maximum diameter of the lump <1.5cm.
6. with enough breast tissue, and enough space from lump to skin.
7. clinically N0 before cryo-ablation.
8. patients is not pregnant and has no plan for pregnancy in 2 years.
9. ECOG level: 0-2
10. serum creatinine≤1.1 mg/dl
11. for patients with double side (left and right side) breast cancer, both side of the tumor should meet the inclusion criteria.
12. patients are accessible for the follow up and mentally healthy.

Exclusion Criteria:

stage 1:

1. < 18 years old
2. male
3. the same side breast of the lump have been treated by surgery or other physical treatment within 3months.
4. benign tumor or tumor in situ or tumor in situ with micro-invasion proved by core needle biopsy. Pathological report is not complete (with the result of ER, PR , HER2, KI67 etc., and FISH report of ERBB2 gene if necessary).
5. image results (including ultrasound, mammography and MR image) prove the lump is multi-center, the maximum diameter of the lump ≥2cm.
6. image results (including ultrasound, mammography) prove calcium region ≥ 5mm
7. lump can not be clearly detected by ultrasound. For example, the boundary of tumor is not clear, or the maximum diameter detected by MRI is more than 1.5 times larger than the maximum diameter detected by ultrasound.
8. before the endpoint, patients is treated by other local treatment.
9. ECOG Level >2
10. serum creatinine>1.1 mg/dl
11. patients are not accessible for the follow up and mentally unhealthy.
12. patients are pregnant or lactating, or have plan for pregnancy in 2 years.
13. other situations which make patients not suitable for the trail or cryo-ablation.

stage 2:

1. < 18 years old
2. male
3. the same side breast of the lump have been treated by surgery or other physical treatment within 3months.
4. benign tumor or tumor in situ or tumor in situ with micro-invasion proved by core needle biopsy. Pathological report is not complete (with the result of ER, PR , HER2, KI67 etc., and FISH report of ERBB2 gene if necessary).
5. absolute contraindication for breast conserving surgery.
6. image results (including ultrasound, mammography and MR image) prove the lump is multi-center, the maximum diameter of the lump ≥1.5cm.
7. image results (including ultrasound, mammography) prove calcium region ≥ 5mm
8. lump can not be clearly detected by ultrasound. For example, the boundary of tumor is not clear, or the maximum diameter detected by MRI is more than 1.5 times larger than the maximum diameter detected by ultrasound.
9. NOT clinically N0 before cryo-ablation.
10. patients are treated after neoadjuvant chemotherapy or neoadjuvant endocrine therapy.
11. patients with advanced breast cancer or other type of cancers.
12. with BRCA1/2 mutation
13. before the endpoint, patients is treated by other local treatment.
14. ECOG Level >2
15. serum creatinine>1.1 mg/dl
16. can not finish the radiotherapy afterwards or with contraindication of radiotherapy
17. patients are not accessible for the follow up and mentally unhealthy.
18. patients are pregnant or lactating, or have plan for pregnancy in 2 years.
19. other situations which make patients not suitable for the trail or cryo-ablation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Stage 1: Effectiveness of cryo-ablation | 1 month
  In the first stage, patients will receive traditional surgery 1month after the cryo-ablation. After the traditional surgery (mastectomy or breast conserving surgery), the pathological report will show whether there is tumor tissue left in the breast tissue. If there is no tumor left in breast, cryo-ablation is effective in eliminating the tumor. Otherwise, cryo-ablation is ineffective.
Stage 2: LRFS(local-regional free survival) | 5 years
  In the second stage, 5-year local-regional free survival will be evaluated for patients with the treatment of cryo-ablation and traditional surgery is spared.
Stage 2: Effectiveness of cryo-ablation (3 months after cryo-ablation) | 3 month
  In the second stage, patients will receive muti-point core needle biopsy (which collect multi-point tissue from the region which was once the tumor region, as reported by MRI or ultrasound) 3months after the cryo-ablation. After the multi-point core needle biopsy, the pathological report will show whether there there is tumor tissue left in the breast tissue. If there is no tumor left in breast, cryo-ablation is effective in eliminating the tumor. Otherwise, cryo-ablation is ineffective.

SECONDARY OUTCOMES:
Stage 1: instant success rate | 3 minutes
  Instant success rate will be evaluated instantly by the surgeon after the cryo-ablation, by his/her own judgement and ultrasound image.
Stage 1: negative predictive value of ultrasound | 14 days and 28 days
  In the first stage, ultrasound will be conducted twice on day 14 and day 28 after the cryo-ablation (16 or 2 days before the traditional surgery). Negative predictive value of ultrasound will be calculated according to the pathological report after the traditional surgery in day 30. Negative predictive value = number of the patients who is pathologically negative AND ultrasound-negative/ number of patients who is ultrasound-negative
Stage 1: adverse events | 1 month
  Short-term safety of cryo-ablation after the treatment
Stage 2: instant success rate | 3 minutes
  Instant success rate will be evaluated instantly by the surgeon after the cryo-ablation, by his/her own judgement and ultrasound image.
Stage 2: shrinking rate | 5 years
  Comparing with the baseline tumor size, shrinking rate of the lump will be calculated in 3 months, 6 months, 12 months, 18 months, 2 years, 3 years, 4 years, 5 years after cryo-ablation. The size of the lump will be evaluated by MR image.
Stage 2: adverse events | 5 years
  Short-term and long-term safety of cryo-ablation after the treatment
Stage 2: breast self evaluation | 5 years
  breast self evaluation for patients with cryo-ablation and for whom traditional surgery is spared, as assessed by BREAST Q© index. The BREAST-Q has a modular, procedure-specific structure with scales that evaluate both satisfaction and quality of life. Psychometric evaluation reveals high reliability, validity and responsiveness to surgical intervention across all scales. Breast Q is composed of aesthetical and emotional modules, and each score ranges from 1 to 4 points (higher values represent a better self evaluation). By comparing the sum of the score in different modules before and after the surgery, Breast Q can help to facilitate a self evaluation for breast cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Min Shao, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No